CLINICAL TRIAL: NCT05864924
Title: A Phase 1 Study Evaluating the Safety and Efficacy of BRG01 in Subjects With Relapsed/Metastatic EBV-positive Nasopharyngeal Carcinoma
Brief Title: A Phase 1 Study of BRG01 in Subjects With Relapsed/Metastatic Epstein-Barr Virus (EBV)-Positive Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioSyngen Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOSG-BRG-01
Record Dates: First submitted 2023-04-27; First posted 2023-05-18 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-04

CONDITIONS: EBV-positive Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BRG01 injection (Experimental): Intravenous infusion
  Interventions: Biological: Cohort A: 3.0x10^6 CAR-T cells/kg; Biological: Cohort B: 9.0x10^6CAR-T cells/kg; Biological: Cohort C:1.5x10^7 CAR-T cells /kg

INTERVENTIONS:
Biological: Cohort A: 3.0x10^6 CAR-T cells/kg — Intravenous infusion
Biological: Cohort B: 9.0x10^6CAR-T cells/kg — Intravenous infusion
Biological: Cohort C:1.5x10^7 CAR-T cells /kg — Intravenous infusion

SUMMARY:
Phase 1 study evaluating the safety and efficacy of BRG01 in subjects with relapsed/ metastatic EBV-positive nasopharyngeal carcinoma (NPC).

BRG01 is a Chimeric Antigen Receptor T-Cell therapy targetting on the specific protein of EBV, which is expressed on the EBV associated cancer cells.

This study adopts the traditional "3+3" dose escalation design. Approximately12~18 EBV+ NPC subjects will be enrolled to evaluate the safety of BRG01. An internal safety review team (SRT) will review the safety data and make recommendations on further study conduct and progression to subsequential cohorts.

Subjects will be enrolled into 3 cohorts of different doses, designated as cohort A, B and C.Cohort A: 3.0x10^6 CAR-T cells/kg,3 subjects, Cohort B: 9.0x10^6 CAR-T cells/kg,3 subjects, and Cohort C:1.5x10^7 CAR-T cells /kg, 6 subjects,respectively.

Subjects in each cohort will follow the same treatment schedule and procedural requirements.

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the safety and efficacy of BRG01.

Secondary Objectives:

1. To evaluate the pharmacokinetics (PK)，pharmacodynamics (PD) and immunogenicity of BRG01.
2. To evaluate the preliminary efficacy of BRG01 in patients with relapsed/metastatic EBV+ NPC.

Exploratory Objectives:

1. To explore the correlation between the proliferation and persistence of BRG01 cells in vivo and the efficacy.
2. To explore the correlation between target expression level in tumor tissue with the safety and efficacy.
3. To explore the correlation between plasma EBV DNA level with safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed nasopharyngeal carcinoma;
2. Be able to understand this study and have signed the informed consent;
3. Age >18 years old, <75 years old;
4. Expected survival period ≥3 months;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
6. Epstein-Barr virus Encoded RNAs (EBER) positive in tumor tissue detected by in situ hybridization (ISH or FISH):
7. By immunohistochemistry (IHC), the target in the pathological sample of the tumor tissue is positive and >20%;
8. According to RECIST v1.1, there is at least one measurable lesion;
9. Patients must have failed to response at least 2 lines of the standard therapies recommended by local NPC guidance, and without other therapy available.
10. Venous access for apheresis or blood collection can be established, without contraindications for leukapheresis;
11. Having adequate organ and bone marrow function, as defined below:

Complete Blood Count Neutrophils (NEUT#) ≥1.0x10^9/L; Platelet (PLT) ≥80x10^9/L; Hemoglobin ≥90g/L; Liver function: Without No liver metastasis Aspartate aminotransferase (AST) ≤2.5 x Upper Limit of Normal (ULN); Alanine aminotransferase (ALT) ≤2.5 x ULN; Total bilirubin (TBIL) ≤1.5 x ULN; Liver Function: With liver metastasis Aspartate aminotransferase (AST) ≤5 x ULN; Alanine aminotransferase (ALT) ≤5 x ULN; Liver Function: With liver metastasis or Gilbert syndrome; Total bilirubin (TBIL) ≤2 x ULN; Creatinine Clearance Rate (CCR) ≥ 50 mL/min; International Normalized Ratio (INR) ≤1.5xULN; Activated partial thromboplastin time (APTT) ≤1.5xULN;

12. During the study period and within 6 months after the end of administration, the subjects of childbearing potential (whether male or female) must use effective medical contraceptive measures For female subjects of childbearing age, a pregnancy test must be performed within 72 hours before cell infusion, and the result is negative.

-

Exclusion Criteria:

1. Known or suspected being allergy to any of the agents used in this study.
2. Previously received anti-tumor treatments, including other anti-tumor investigational drugs, chemotherapy, immunotherapy, biological agents, hormone therapy, radiation therapy (except local radiation therapy for pain relief), etc., the treatment related toxicity not recovered to baseline or CTCAE≤0~1.
3. Received adoptive cellular immunotherapy (including CAR-T cells and T Cell Receptor-T cells (TCR-T)) within 6months.
4. Confirmed central nervous system metastasis.
5. Confirmed extensive liver metastasis (the tumor volume is estimated to be≥50% of the total liver volume imaging).
6. Clinically significant active infections (e.g. Simple Urinary Tract Infection (UTl), bacterial pharyngitis are allowed) or currently receiving IV antibiotics or have received IV antibiotics with in 14 days prior to enrollment(Prophylaxis antibiotics, antivirals and antifungals are permitted);
7. HBsAg positive and Hepatitis B Virus (HBV) DNA copy number positive (quantitative detection ≥1000cps/ml), Hepatitis C Virus (HCV) antibody positive and HCV RNA positive, or HIV positive.
8. History of autoimmune diseases (e.g, primary immunodeficiency, inflammatory bowel disease. idiopathic thrombocytopenic purpura, systemic lupus erythematosus, autologous hemolytic anemia, rheumatoid arthritis, etc.).
9. The following diseases have not been resolved to CTCAE grade 0-1, 7 days before the conditioning chemotherapy, including: dyspnea, diarrhea, acute or chronic pancreatitis.
10. New York Heart Association (NYHA) class 3 or 4.
11. Symptoms and sign of cardiovascular diseases, e.g., cardiovascular ischemia, arrhythmias, and heart failure.
12. Symptoms and signs of cerebrovascular accidents.
13. History of other malignant tumors that cannot be cured within 3 years, except for cervical cancer in situ or skin basal cell carcinoma, and other malignant tumors with a disease-free survival period of more than 5 years.
14. Current or expected need for long-term systemic corticosteroid therapy. Note: Topical and inhaled corticosteroids in standard doses and physiologic replacement for subjects with adrenal insufficiency are allowed. Doses of corticosteroids of greater than or equal to 5 mg/day of prednisone or equivalent doses of other corticosteroids are not allowed.
15. Subjects of both genders who are not willing to practice birth control from the time of consent through 6 months after the completion.-
16. Subjects have experienced major surgery or severe trauma within 4 weeks before enrollment or are expected to undergo major surgery during the study period.
17. Combined with graft versus host disease (GVHD).-
18. Women of child-bearing potential who are pregnant or breastfeeding at the screening. Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential.
19. Patients with confirmed history of neurological or psychotic disorders, including epilepsy, seizure, dementia.
20. Any other condition that, in the discretion of the investigator, will make subjects exposed to unnecessary risks or not compliance to participation in this clinical study.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | From the infusion (Day 0) to Day 28
  Incidence of adverse events defined as Dose-Limiting Toxicity (DLT).
Maximum tolerated dose | From the infusion (Day 0) to Day 28
  The maximum CAR-T dose that can be tolerated in the study.
AE, SAE, AESI, CRS, ICANS, TEAE | The day of leukapheresis to 3 months after infusion
  The incidence of adverse events (AE), serious adverse events (SAE), adverse events of special interest (AESI), cytokine release syndrome (CRS) immune cell associated neurotoxicity syndrome (ICANS) and treatment-emergent adverse events (TEAE).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No